CLINICAL TRIAL: NCT03036618
Title: Effects of Quinoa Consumption on Markers of Cardiovascular Risk and Gastrointestinal Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUHEALTH-LL01-Quinoa
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Change in Fasting Plasma LDL-cholesterol Concentration After the Consumption of Quinoa
Keywords: BMI; Blood Cholesterol; Glucose; Insulin; Gut health
MeSH Terms: conditions — Insulin Resistance | interventions — chenopodin protein, Chenopodium quinoa; Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wheat (Placebo Comparator): Test wheat bread roll (approximately 160g weight) without quinoa.
  Interventions: Dietary Supplement: Wheat
- Quinoa (Experimental): Test wheat bread roll (approximately 160g weight) delivering 20 g quinoa consumed per day.
  Interventions: Dietary Supplement: Quinoa

INTERVENTIONS:
Dietary Supplement: Quinoa — Test wheat bread roll (approximately 160g weight) delivering 20 g quinoa consumed per day.
  Arms: Quinoa
Dietary Supplement: Wheat — Test wheat bread roll (approximately 160g weight) without quinoa.
  Arms: Wheat

SUMMARY:
Quinoa is possible alternative to wheat, corn and rice due to its high nutritional value and possible properties against cardiovascular diseases and for improving gut health. There are some animal studies to suggest that some important class of compounds like fibre, antioxidants and protein, found naturally in quinoa, have beneficial effects against markers of cardiovascular diseases. However, the effects of quinoa on humans has rarely been investigated. This study will investigate the effects of daily consumption of quinoa for four weeks on markers of cardiovascular risk, including blood cholesterol and resting blood pressure, and on gut health in a randomised cross-over study design.

DETAILED DESCRIPTION:
Quinoa is a possible alternative to wheat, corn and rice due to its high nutritional value and possible properties against cardiovascular diseases. There are some animal studies which suggest that quinoa has beneficial effects against markers of cardiovascular diseases, particularly blood lipid profile. The grain has a unique nutritional profile, with high fibre levels and a wide range of phytochemicals which may influence gut bacteria and improve gastrointestinal health.

However, the effects of quinoa on humans has rarely been investigated with just two small interventions published. These studies also showed an improvement in blood lipid profile after consuming quinoa daily. There have been no studies which have investigated the effects of quinoa on gut bacteria and gastrointestinal health. Therefore, this human dietary intervention study aims to determine the effects of quinoa consumption on markers of cardiovascular diseases, the gut microbiome and gastrointestinal health.

The study is a randomized cross-over designed dietary intervention study with 4-week study periods separated by a 4-week wash-out period. The treatment will be the daily consumption of a test bread roll containing quinoa to deliver 20g quinoa per day (one roll per day). The control will be the same amount of a refined wheat roll. Markers of cardiovascular disease risk, including fasting blood lipid profile, plasma glucose and insulin concentration, resting blood pressure will be compared at the beginning and end of each treatment period. Changes in the numbers and species of gut bacteria, and products of bacterial fermentation will be made in stool samples collected at the beginning and end of each intervention period as indicators of gastrointestinal health.

ELIGIBILITY:
Inclusion Criteria:

1. healthy men >35 years old
2. body mass index >25 kg/m2
3. Non-smokers with no known previous history of cardiovascular disease or type 2 diabetes
4. Not receiving any current medication. Supplement users will be included but will be asked to stop taking supplements for the duration of the study

Exclusion Criteria:

1. Age ≤ 35 or BMI ≤25
2. Smokers
3. Individuals with known or suspected allergy to wheat
4. Individuals with known history of cardiovascular diseases or type 2 diabetes
5. Individuals with recent weight loss (>10%) or planning to lose weight during the study

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-02 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
plasma LDL-cholesterol | Change from post dose after 4 weeks of intervention

SECONDARY OUTCOMES:
BMI | Change from post dose after 4 weeks of intervention
Body fat | Change from post dose after 4 weeks of intervention
Blood pressure | Change from post dose after 4 weeks of intervention
Fasting Blood glucose and insulin | Change from post dose after 4 weeks of intervention
Fasting blood lipid profile | Change from post dose after 4 weeks of intervention
Stool Microbiome profile | Change from post dose after 4 weeks of intervention
short chain fatty acid profile of stool samples | Change from post dose after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chris Seal, Professor, Principal Investigator — Newcastle University
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided